CLINICAL TRIAL: NCT05612139
Title: A Single Center Post-market Clinical Follow-up (PMCF) Observational Study Evaluating the Clinical Performance and the Safety Profile of the JuniOrtho™ Telescopic Intramedullary Nail (JTIN) for the Treatment of Pediatric Patients Suffering From Osteogenesis Imperfecta
Brief Title: Post-market Observational Study on JTIN Telescopic Nail in Osteogenesis Imperfecta Pediatric Patients
Acronym: JTIN
Status: Completed | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_2201
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: nailing; nail; Osteogenesis; pediatric; bone; rare disease; brittle; telescopic
MeSH Terms: conditions — Osteogenesis Imperfecta; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JTIN treated patients: Pediatric patients, older than 18 months, suffering from osteogenesis imperfecta treated with JTIN telescopic nail
  Interventions: Device: JTIN implantation surgery

INTERVENTIONS:
Device: JTIN implantation surgery — The JTIN is a self-extending intramedullary nail (telescopic rod) designed to provide fixation of femoral and/or tibial fractures, osteotomies, malunions and non-unions. The design of the JTIN includes a female and a male component, which are anchored to the proximal cortex and distal epiphysis through screw-type fixation. These two components slide from each other, allowing for extension of the JTIN as the bone structures remodel and patient growth occurs.

SUMMARY:
This study has been planned as part of the Orthofix Srl post-market active surveillance plan for the collection of data on both the clinical performance and the safety profile of the JTIN.

The rationale of the proposed study is to update and support the pre-market clinical evaluation of the JTIN with Real World Evidence clinical data in a real-life surgical setting, in order to confirm the benefit/risk ratio of this medical device and to keep the CE mark under Medical Device Regulation (MDR) requirements. One selected site, experienced in the treatment of pediatric patients with OI, where the usage of JTIN is already part of the normal clinical practice, will participate in this study.

DETAILED DESCRIPTION:
One selected site, experienced in the treatment of pediatric patients with OI, where the usage of JTIN is already part of the normal clinical practice, will participate in this study. Investigator will screen patients treated (or planned to be treated) with JTIN to verify inclusion and exclusion criteria, to achieve the enrollment of 25 cases. With lost to follow-up percentage estimated at 20%, this will lead to a total of 20 evaluable cases, i.e. 20 implanted JTIN (some patients may contribute for more than one implant). Patients are prospectively and retrospectively enrolled in the study: they may have undergone JTIN implantation from the 1st of January 2022.

Enrolled patients, since this study is non-interventional and observational, will follow the standard medical practice of the site: no requirements regarding the treatment of patients will be imposed on the site or Principal Investigator and the Sponsor will not in any manner influence the treatment decisions. Data of enrolled subjects will be collected for this study up to 1 year from surgery.

The hospital standard care usually, but not exclusively, includes: surgery, discharge and plaster removal visits, and then 3 other follow up visits up to 1 year from surgery (see "Visits and Assessments Schedule"). Visits frequency is estimated as average of the site normal clinical practice, actual visit timing for each patient will be performed according to investigators and hospital staff evaluation.

The patient data will be systematically collected by the investigator in eCRF.

ELIGIBILITY:
Inclusion Criteria:

* is in pediatric age (> 18 month and < 18 years) at the time of surgery;
* is skeletally immature;
* has a diagnosis for OI;
* has a regular indication for surgical intervention with JTIN to treat femoral and/or tibial fractures, osteotomies, malunions and non-unions;
* patient and/or legal representative is duly informed and doesn't oppose to participation.

Exclusion Criteria:

* has a medical condition that is a contraindication according to the manufacturer's instruction for use;
* has any conditions that in the Investigator's opinion may interfere with the study execution or due to which the patient should not participate for safety reasons;
* requires the application of, or has already in-situ the application of concomitant devices that cannot be safely removed (except for permitted concomitant devices paragraph);
* is participating in other clinical trials or has taken part in any clinical study in the last 3 months with exception of analytical trials on genetics study related to OI (i.e. studies that do not include an investigational treatment for the patient such as new drugs or other medical devices);
* is likely to be lost to follow up, according to investigator's opinion.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients older than 18 months suffering from osteogenesis imperfecta.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zagorka Pejin, MD, Principal Investigator — Necker-Enfants Malades Hospital
Locations (1):
- Necker-Enfants Malades Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azzam KA, Rush ET, Burke BR, Nabower AM, Esposito PW. Mid-term Results of Femoral and Tibial Osteotomies and Fassier-Duval Nailing in Children With Osteogenesis Imperfecta. J Pediatr Orthop. 2018 Jul;38(6):331-336. doi: 10.1097/BPO.0000000000000824. PMID 27379783
- [Background] Birke O, Davies N, Latimer M, Little DG, Bellemore M. Experience with the Fassier-Duval telescopic rod: first 24 consecutive cases with a minimum of 1-year follow-up. J Pediatr Orthop. 2011 Jun;31(4):458-64. doi: 10.1097/BPO.0b013e31821bfb50. PMID 21572286
- [Background] Novacheck TF, Stout JL, Tervo R. Reliability and validity of the Gillette Functional Assessment Questionnaire as an outcome measure in children with walking disabilities. J Pediatr Orthop. 2000 Jan-Feb;20(1):75-81. PMID 10641694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient information and the collection of the non-opposition form could also be carried out after the patient's treatment, as the study is entirely observational and allows for the inclusion of retrospective patients. This was the case for all patients included in the study: all had undergone surgery with JTIN before the study began and were therefore informed about the study after their treatment.
Units Other Than Participants: implants (i.e. procedures)
Period: Overall Study
Arm/Group | JTIN Treated Patients
Started | 14; 25 implants (i.e. procedures)
Completed | 14; 25 implants (i.e. procedures)
Not Completed | 0; 0 implants (i.e. procedures)

BASELINE CHARACTERISTICS:
Population: The study was performed in 14 pediatric patients who had a regular indication for surgical intervention with JTIN and in this document are reported the results obtained in 25 surgical procedures.
Arm/Group | JTIN Treated Patients
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at surgery | 5.4 (3.0)
  Age at study inclusion | 7.5 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Procedures With at Least One Serious/Not Serious Adverse Event Certainly or Possibly Related to JTIN
Description: The primary endpoint is measured to evaluate the clinical safety profile of JTIN within the scope of its intended purpose.
Time Frame: 1 year
Population: A total of 25 implants where analyzed on 14 recruited patients, therefore the population included in the final analysis is 25 implants and 14 patients.
Measure: Number (95% Confidence Interval); unit: percentage of procedures
Units Other Than Participants: Implants (i.e. procedures)
Arm/Group | JTIN Treated Patients
Number analyzed (Participants) | 14
Number analyzed (Implants (i.e. procedures)) | 25
percentage of procedures | 4.0 [0.1 to 20.4]

2. Secondary Outcome: Implant Survival Rate: Percentage of Not Exchanged Nails
Description: This endpoint measures how many nails, in percentage, remains functional in the patient without requiring surgical replacement. Specifically, it represents the proportion of implanted nails that do not need to be exchanged during the follow-up period for any reason. A higher implant survival rate indicates better durability, safety for patients and clinical performance. This endpoint is measured to evaluate the clinical safety of JTIN.
Time Frame: 1 year
Population: A total of 25 implants for 14 patients have been recruited, therefore the population included in the final analysis is 25 implants and 14 patients.
Measure: Number (95% Confidence Interval); unit: percentage of not exchanged nails
Units Other Than Participants: Implants (i.e. procedures)
Arm/Group | JTIN Treated Patients
Number analyzed (Participants) | 14
Number analyzed (Implants (i.e. procedures)) | 25
percentage of not exchanged nails | 100.0 [86.3 to 100.0]

3. Secondary Outcome: Percentage of Procedures With Bone Union Achievement
Description: This endpoint is measured to evaluate the clinical performance of JTIN.
Time Frame: 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of procedures
Units Other Than Participants: Implants (i.e. procedures)
Arm/Group | JTIN Treated Patients
Number analyzed (Participants) | 14
Number analyzed (Implants (i.e. procedures)) | 25
percentage of procedures | 100.0 [86.3 to 100.0]

4. Secondary Outcome: Post-treatment Fracture-free Survival Rate
Description: This endpoint is measured to evaluate the clinical performance of JTIN.
  This endpoint is described with the percentage of patients that experienced a fracture of the JTIN-treated bone during the specified time frame.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | JTIN Treated Patients
Number analyzed (Participants) | 14
percentage of patients | 35.7 [12.8 to 64.9]

ADVERSE EVENTS:
Time Frame: The Adverse Event where collected from surgery to last time point indicated in the protocol (1 year + 1 month, total of 13 months post-surgery)
Description: The investigator will follow the standard clinical practice to record data in the medical file. In addition to the above-mentioned requirements, the investigator will also record the AEs and MDDs in the eCRF. For both cases the investigator, when reporting the event in the eCRF will describe: date of the event; treatment; resolution; whether or not it is Serious and whether or not it is related to the use of the investigational device and the related procedure.
Arm/Group | JTIN Treated Patients
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTIN Treated Patients (N=14)
Non-union, delayed union or malunion (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone fracture during or after treatment (Injury, poisoning and procedural complications) | 7 (7)
Migration of the device (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTIN Treated Patients (N=14)
Bone fracture during or after treatment (Injury, poisoning and procedural complications) | 10 (17)
Pain, discomfort or abnormal sensations due to the presence of the device (Injury, poisoning and procedural complications) | 2 (2)
Residual deformities, persistence or recurrence of the initial condition subject to treatment (Musculoskeletal and connective tissue disorders) | 1 (1)
Stiffness at surgery site (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor recognizes co-authors' right to publish non-commercial study results after the sponsor's first publication. Co-authors must submit manuscripts or abstracts to the sponsor at least 30 days before publication; the sponsor will provide comments within 15 working days. The sponsor and investigator may also publish results and submit data to regulatory authorities. The sponsor's identity and contribution must be disclosed in all publications.

DOCUMENTS (2):
  • Study Protocol (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT05612139/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT05612139/SAP_001.pdf